CLINICAL TRIAL: NCT02893358
Title: Antihypertensive Treatment in Masked Hypertension for Target Organ Protection (ANTI-MASK)
Brief Title: Antihypertensive Treatment in Masked Hypertension
Acronym: ANTI-MASK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yan Li (Other)
Responsible Party: Sponsor-Investigator, Yan Li, Professor, Doctor of Medicine, Doctor of Philosophy, Shanghai Institute of Hypertension
Organization: Shanghai Institute of Hypertension (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANTI-MASK20160830
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Masked Hypertension
Keywords: Allisartan Isoproxil; left ventricular hypertrophy; large arterial stiffness; microalbuminuria
MeSH Terms: conditions — Masked Hypertension; Hypertrophy, Left Ventricular | interventions — allisartan isoproxil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment (Active Comparator): Treatment will be started with allisartan isoproxil 80mg once daily taken in the morning during 8:00-9:00. After 2 months, to achieve the target BP (24h BP<130/80 mmHg, and daytime BP <135/85 mmHg, and nighttime BP <120/70 mmHg), allisartan isoproxil may be doubled to 160mg once a day. If necessary, amlodipine 2.5mg may be combined with allisartan Isoproxil.
  Interventions: Drug: Allisartan Isoproxil
- Placebo (Placebo Comparator): Placebo tablets are identical to the active study drugs, with a similar schedule of administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Allisartan Isoproxil — Allisartan Isoproxil 80mg once daily taken in the morning during 8:00-9:00. To achieve the target blood pressure allisartan isoproxil may be doubled to 160mg once a day. If necessary, amlodipine 2.5mg may be combined with allisartan isoproxil. Duration: 12 months.
  Arms: Active treatment
Drug: Placebo — Corresponding placebo once daily taken in the morning during 8:00-9:00. Duration: 12 months.
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to estimate the target organ protection after 12 months of antihypertensive treatment in masked hypertension patients with at least one kind of target organ damage (left ventricular hypertrophy, large arterial stiffness and microalbuminuria). Improvement was defined as the relevant parameter back to normal or declined at least 20%.

The secondary objectives include: blood pressure lowering effect, target organ damage parameters improvement, and the incidence rate of all cause death and cardiovascular events (stroke and myocardia infraction).

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-70 years old
2. Masked hypertension patients, defined as clinic BP<140/90 mmHg, while 24h ambulatory BP ≥130/80 mmHg and (or) daytime BP ≥135/85 mmHg and (or) nighttime BP ≥120/70 mmHg
3. Combined with at least one kind of target organ damage: left ventricular hypertrophy (Cornell voltage combination ≥2440mm·ms or Sokolow-Lyon index ≥4.0mv for male and 3.5mv for female), large arterial stiffness (brachial-ankle pulse wave velocity ≥1400cm/s) and microalbuminuria (twice random urine microalbuminuria/creatinine ratio ≥2.5mg/mmol for male and 3.5mg/mmol for female).
4. Didn't use any anti-hypertension drugs within 2 weeks
5. Be willing to participate in the trials and able to finish clinic visits

Exclusion Criteria:

1. Under antihypertensive treatment
2. Secondary hypertension
3. Taking other medications that may influence BP
4. Sleep apnea syndrome
5. Diabetes combined with microalbuminuria
6. Renal parenchymal disease, such as chronic nephritis, polycystic kidney
7. Occurrence of coronary heart disease, myocardial infraction or stroke within 6 months
8. Structural heart disease, such as hypertrophic cardiomyopathy, dilated cardiomyopathy
9. Alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin (TBL) upper the twice of normal range, serum creatinine (Scr)≥2.0mg/dl, plasma hypokalemia≥5.5mmol/L,
10. Patients have contraindications to angiotensin receptor blockers (ARBs)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Improvement rate of target organ damage (left ventricular hypertrophy, large arterial stiffness and microalbuminuria) | 1 year
  Improvement was defined as the relevant parameters (Cornell voltage combination, Sokolow-Lyon index, microalbuminuria/creatinine ratio, brachial-ankle pulse wave velocity) back to normal or declined at least 20%.

SECONDARY OUTCOMES:
24h ambulatory blood pressure | 1 year
electrocardiogram | 1 year
  calculating Cornell voltage combination and Sokolow-Lyon index
microalbuminuria/creatinine ratio | 1 year
brachial-ankle pulse wave velocity | 1 year
incidence rate of all cause death and cardiovascular events (stroke and myocardia infraction) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang JF, Zhang DY, An DW, Li MX, Liu CY, Feng YQ, Zheng QD, Chen X, Staessen JA, Wang JG, Li Y; ANTI-MASK Investigators. Efficacy of antihypertensive treatment for target organ protection in patients with masked hypertension (ANTI-MASK): a multicentre, double-blind, placebo-controlled trial. EClinicalMedicine. 2024 Jul 18;74:102736. doi: 10.1016/j.eclinm.2024.102736. eCollection 2024 Aug. PMID 39091669